CLINICAL TRIAL: NCT07130214
Title: The Effect of Genetic Polymorphisms on the Success of Vital Pulp Therapy
Status: Active, not recruiting | Type: Observational
Sponsor: Ataturk University (Other)
Collaborators: Health Institutes of Turkey (Other Government)
Responsible Party: Principal Investigator, ertuğrul karataş, Professor, Ataturk University
Other Study IDs: B.30.2.ATA.0.01.00/242; 48446 (Other: TUSEB)
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Pulp Exposure, Dental; Pulp Disease, Dental; Pulp Caping; Pulpitis; Pulpitis - Irreversible; Pulpal Inflammation
Keywords: Biodentine; Pulp Capping; SNP
MeSH Terms: conditions — Dental Pulp Exposure; Dental Pulp Diseases; Pulpitis | interventions — tricalcium silicate; Pemetrexed; Healthco pulp capping material

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Patient indicated with pulp capping: In the planned project,vital pulp therapy will be applied to teeth diagnosed with reversible or irreversible pulpitis,showing a positive response to vitality tests and no periapical radiolucency.
  Interventions: Drug: Biodentine

INTERVENTIONS:
Drug: Biodentine — Biodentine is used in the treatment of existing dentin damage thanks to active bio-silicate technology.
  Other Names: MTA; Pulp Capping Material

SUMMARY:
This study employs saliva-based DNA analysis to investigate the effect of genetic polymorphisms, particularly SNPs in MMP, TIMP, TNF-α, and BMP genes, on the success of vital pulp therapy in permanent teeth with pulpitis, assessed through clinical follow-up.

DETAILED DESCRIPTION:
The treatment choice following pulp exposure due to dental caries in permanent mature teeth is still a topic of debate today.Vital pulp therapy is recommended in teeth with reversible or irreversible pulpitis which do not show periapical inflammation as it helps preserve the pulp's defense mechanism and facilitates new dentin formation.The success of vital pulp therapy depends on various factors such as age,the size of the exposed area,the amount of remaining tooth and response to vitality tests.It is known that the genetic makeup of patients can influence the success of vital pulp therapy.These genetic differences may arise from polymorphisms occurring in an individual's DNA sequence at a frequency of 1% or higher.Single nucleotide polymorphisms(SNPs)are considered the most common type of polymorphism and are thought to occur every 1000 base pairs in the human genome.Matrix metalloproteinases(MMPs),tissue inhibitors of metalloproteinases(TIMPs),tumor necrosis factor-α(TNF-α),bone morphogenic proteins(BMPs)which affect inflammation pathways and tissue remodeling,can also influence the success of this treatment.MMPs are associated with the degree of inflammation and the destruction of pulp tissues.They are crucial in the formation of the dentin matrix and secondary dentin and also immune response development.They are inhibited by TIMPs which are endogenously secreted. Polymorphisms in the MMP and TIMP genes increase the susceptibility of patients to pulp tissue destruction. MMP-9 facilitates tissue degradation in inflamed pulp tissue.TNF-α is a pro-inflammatory cytokine.The elevation of TNF-α levels in the pulp triggers inflammatory reactions by stimulating pulp cells to produce MMPs.BMPs promote the conversion of osteoprogenitor cells into osteoblasts.Specifically,BMP-4 factor initiates dentin formation.Therefore,it is likely that SNPs in the genes coding for these inflammatory mediators and growth factors can influence the success of vital pulp therapy.In the planned project,vital pulp therapy will be applied to teeth diagnosed with reversible or irreversible pulpitis,showing a positive response to vitality tests and no periapical radiolucency.Saliva samples will be collected from the included patients in Eppendorf tubes.After local anesthesia,the tooth will be isolated with a rubberdam and the decayed tissue will be removed until it reaches hard healthy dentin.The bleeding from the exposed pulp will be controlled for 30 seconds with a cotton pellet soaked in 2.5% NaOCl solution.After irrigation with sterile saline, the exposed area will be capped with a calcium silicate-based material called Biodentine(Septodont,France).The material will be sealed with resin-modified glass ionomer cement, and a permanent restoration will be placed.After the procedure,patients will be clinically and radiographically evaluated with a 12-month follow-up.DNA will be isolated from the saliva samples and the relationship between SNPs in the relevant genes and treatment success will be determined.

ELIGIBILITY:
Inclusion Criteria

* permanent teeth diagnosed with reversible pulpitis,
* patients diagnosed with irreversible pulpitis but without apical radiolucency, -teeth responding within normal limits to cold stimuli (using carbon dioxide snow),
* teeth with prolonged response to cold testing, diagnosed with irreversible pulpitis,
* teeth without sensitivity to percussion or chewing tests,
* teeth with bleeding time less than 5 minutes from exposed pulp tissue,
* teeth diagnosed with irreversible pulpitis with bleeding time less than 10 minutes,
* teeth without widening of the periodontal ligament space (Periapical Index [PAI] ≥2),
* teeth with radiographically confirmed deep dentinal caries,
* patients classified as ASA I (American Society of Anesthesiologists Physical Status Classification)

Exclusion Criteria:

* teeth showing negative response to cold testing (using carbon dioxide snow), -teeth showing negative response to electric pulp testing,
* presence of apical radiolucency (PAI > 2),
* presence of condensing apical periodontitis in the relevant tooth,
* teeth with internal or external root resorption,
* teeth with a history of trauma,
* teeth with vertical root fractures,
* evidence of periodontal-endodontic lesion on the day of treatment,
* loss of function (e.g., tooth mobility degree 3),
* presence of swelling related to the treated tooth,
* teeth that cannot be treated with rubber dam isolation,
* patients with compromised immune systems,
* patients who are pregnant at the time of treatment,
* patients who have used antibiotics, bisphosphonates, or statins within the last 4 weeks prior to treatment.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Ataturk University Faculty of Dentistry Endodontics Department
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2025-05-02 (Actual); Primary Completion 2026-05-02 (Estimated); Study Completion 2026-11-02 (Estimated)

PRIMARY OUTCOMES:
DNA Analysis | From enrollment to the end DNA analysis at 18 months
  After treatment, patients will undergo clinical and radiographic evaluations at the 6th and 12th months. Treatments will be considered successful if the patient reports no complaints during follow-up; if clinical examination reveals no hypersensitivity to thermal stimuli, gingival swelling, sinus tract, mobility, or sensitivity to lateral and vertical percussion; and if radiographic examination shows no periradicular changes, root resorption, irregular calcification within the canal, and evidence of a radiopaque dentin bridge formation.After the 12-month follow-up period, the data obtained will be categorized according to patients' genetic profiles (i.e., polymorphism types), and the relationship between vital pulp therapy success and genetic polymorphism will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided